CLINICAL TRIAL: NCT00222638
Title: Randomized Blinded Cross-Over Clinical Trial Investigate the Interactions Between Influenza Vaccination and Oral Anticoagulant Therapy
Brief Title: Influenza Vaccination and Oral Anticoagulant Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Of Perugia (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 04 MICV AI 01
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2005-09-22 (Estimated); Status verified 2005-06

CONDITIONS: Anticoagulants; Influenza Vaccines
Keywords: Oral anticoagulants; Influenza virus; Influenza vaccine; Pharmacological interference
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Drug: Influenza vaccination

SUMMARY:
The purpose of this study is to evaluate INR and INR related index and Warfarin weekly dosage variations after Influenza Vaccination

DETAILED DESCRIPTION:
The pharmacokinetic and the pharmacodynamic interactions and the possible clinical events connected with the simultaneous administration of Oral Anticoagulants (OA) and the influenza virus vaccine were evaluated in several small studies which yielded conflicting results, thus encouraging additional investigations with prospective studies in order to obtain a more consistent evidence about the safety and efficacy of vaccination against influenza virus in patients on OA Treatment.

ELIGIBILITY:
Inclusion Criteria:

* OA Treatment
* Stable anticoagulation (previous two controls in range)
* Presence of indication for Influenza Vaccination
* Life expectancy > 6 months
* Signed Informed consent

Exclusion Criteria:

* Absence of stable anticoagulation
* Absence of indication for Influenza Vaccination
* Life expectancy < 6 months
* Denied Informed Consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-10; Study Completion 2005-05

PRIMARY OUTCOMES:
1.Variations in INR value and in OAT weekly dosage after IV

SECONDARY OUTCOMES:
1.Efficacy of IV in patients on OAT

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Iorio, Principal Investigator — University Of Perugia; Maria Vecchioli, Principal Investigator — Regional Sanitary Agency (ASL2-Perugia); Anna Maria Iorio, Principal Investigator — Institute of Virology - University of Perugia
Locations (1):
- University of Perugia, Perugia, Perugia, Italy

REFERENCES:
- [Derived] Iorio A, Basileo M, Marcucci M, Guercini F, Camilloni B, Paccamiccio E, Vecchioli M, Iorio AM. Influenza vaccination and vitamin K antagonist treatment: a placebo-controlled, randomized, double-blind crossover study. Arch Intern Med. 2010 Apr 12;170(7):609-16. doi: 10.1001/archinternmed.2010.49. PMID 20386004